CLINICAL TRIAL: NCT06108934
Title: A Prospective, Pre-market, Multi-center Evaluation of the Clinical Outcomes of the Insignia Hip Stem in Total Hip Arthroplasty (THA)
Brief Title: A Prospective, Pre-market, Multi-center Study of Insignia Hip Stem in THA to Determine Implant Survivorship and PROMS.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Stryker South Pacific (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Insignia-23
Record Dates: First submitted 2023-10-18; First posted 2023-10-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Arthritis (E.G., Degenerative Joint Disease (DJD), Osteoarthritis, and Rheumatoid Arthritis (RA))
MeSH Terms: conditions — Arthritis; Joint Diseases; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention group (Experimental): Insignia hip stem study group
  Interventions: Device: Hip stem prosthesis

INTERVENTIONS:
Device: Hip stem prosthesis — The Insignia hip stem prosthesis will be used in cementless total hip replacement surgery (THA). The surgery typically takes approximately two hours. All study participants will receive the Insignia hip stem and compatible components. Experienced Orthopaedic Surgeons trained in THA will perform the surgeries as per the standard surgical technique guide for this prosthesis.

SUMMARY:
The purpose of this study is to evaluate the survivorship (revision rates) and patient reported outcomes (PROMs) following implantation of the Insignia hip stem in patients undergoing cementless total hip replacement surgery compared to currently available stems used for the same type of surgery.

It is hypothesised the 2-year survivorship of the Insignia stem is noninferior to the benchmark survivorship of similar stems used in the same type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed the study specific, Human Research Ethics Committee (HREC) approved, Patient Information Consent Form for the use of the study device
* Primary non-inflammatory degenerative joint disease (including osteoarthritis or avascular necrosis) and/or rheumatoid arthritis
* The patient is a candidate for a primary cementless THA.
* Patients who are informed of the conditions of the study and are willing to participate for the length of the prescribed follow-up period.

Exclusion Criteria:

* Active or suspected latent infection in or about the affected hip joint and the time of study device implantation.
* Any mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure or complications in post-operative care.
* Has bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* Is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. >30 days.)
* Requires revision THA or hip fusion to the affected joint.
* Has known sensitivity to device materials.
* Any involvement in an active Workers' Compensation investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship | 2 years post-operatively
  Implant survivorship using cumulative percent revision (CPR) of the Insignia hip stem, for any reason.

SECONDARY OUTCOMES:
Oxford Hip Score | Pre-operatively and 6 months, 12 months and 2 years post-operatively
  Performance of the Insignia hip stem using Oxford Hip Score (OHS) in the intervention group
Hip Disability and Osteoarthritis Outcome Score (HOOS-12). | Pre-operatively and 6 months, 12 months and 2 years post-operatively
  Function, pain and satisfaction in the intervention group using the Hip Disability and Osteoarthritis Outcome Score mid-version (HOOS-12). This is a composite measure.
EQ-5D-5L | Pre-operatively and 6 months, 12 months and 2 years post-operatively
  Function, pain and satisfaction in the intervention group using EQ-5D-5L domains and EQ (Visual analogue scale) VAS. This is a composite measure.
Hip and lower back pain VAS | Pre-operatively and 6 months, 12 months and 2 years post-operatively
  Hip and lower back pain in the intervention group using a VAS. This is a composite measure.
Forgotten Joint Score (FJS) | Pre-operatively and 6 months, 12 months and 2 years post-operatively
  Function, pain and satisfaction in the intervention group using Forgotten Joint Score (FJS). This is a composite measure.
Complications | Collected as they arise post-operatively. Reported as number within 6 months, 12 months and 2 years post-operatively.
  Post-operative complications when the Insignia Hip Stem is used in THA in the intervention group..
Mortality | 1 and 2 years post-operatively
  Mortality in the intervention group
CPR for stem loosening | 2 years post-operatively
  CPR of the Insignia Hip Stem for stem loosening in the intervention group
Femoral fracture | 2 years post-operatively
  Insignia Hip Stem device-related femoral fracture in the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Clark, MD, Principal Investigator — Perth Hip and Knee
Locations (1):
- St John of God Subiaco Hospital, Subiaco, Western Australia, Australia